CLINICAL TRIAL: NCT00825188
Title: Investigation of Reduction of Blood Pressure and Metabolic Rate in Obese Hypertensive Patients Using Eplerenone: Implications for Treatment of Hypertension and Heart Failure
Brief Title: A Study of the Effects of Eplerenone and Amlodipine on Blood Pressure and Basal Metabolic Rate in Obese Hypertensives
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding to complete was inadequate
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Marion Wofford, Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0035
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2014-03

CONDITIONS: Obesity; Hypertension
MeSH Terms: conditions — Obesity; Hypertension | interventions — Eplerenone; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- eplerenone (Active Comparator)
  Interventions: Drug: eplerenone, amlodipine; Drug: eplerenone; Drug: amlodipine
- amlodipine (Active Comparator): Amlodipine 5-10mg daily times 8 weeks
  Interventions: Drug: eplerenone, amlodipine; Drug: eplerenone; Drug: amlodipine

INTERVENTIONS:
Drug: eplerenone, amlodipine — Eplerenone 25mm qd versus amlodipine 5mg qd x 4weeks the Eplerenone 50mg qd versus amlodipine 10mg qd x 4weeks
  Other Names: Inspra; Norvasc
Drug: eplerenone — Eplerenone 25-50mg daily x 8 weeks
  Other Names: Inspra
  Arms: eplerenone
Drug: eplerenone — eplerenone 25- 50 mg daily for 8 weeks
  Other Names: Inspra; Norvasc
Drug: amlodipine — amlodipine 5-10mg daily for 8 weeks
  Other Names: Norvasc

SUMMARY:
Obesity and hypertension are independent risks for congestive heart failure (CHF) and chronic kidney disease. In obesity induced hypertension, the most common cause of human essential hypertension, the potential importance of mineralocorticoid receptor blockade has not been widely investigated. We propose to test the hypothesis that eplerenone reduces metabolic demand, improves cardiac function and attenuates glomerular hyperfiltration and microalbuminuria in obese patients. Our specific aims are to assess changes in basal metabolic rate, cardiac and renal function in obese hypertensive subjects treated with eplerenone compared to amlodipine.

DETAILED DESCRIPTION:
The proposed trial will utilize an open label study design. Patients with hypertension and obesity will be recruited. After a 3-week washout period for patients currently on antihypertensive medication, eligible participants will be assigned to receive 25 mg of eplerenone or 5 mg of amlodipine. After a 4 week period on medication, drug will be advanced to 50 mg of eplerenone or 10 mg of amlodipine for an additional 4 weeks.

Protocol Synopsis:

1. Recruit 20 study participants with a systolic blood pressure (SBP) between 140 and 160 mmHg and/or a diastolic blood pressure between 90 and 100 mmHg who also have a body mass index > 30-45. If participants are on antihypertensive treatment, they will undergo a 3-week washout period. The study participants will be identified in the Division of Hypertension.
2. Assign study participants to receive 25 mg of eplerenone or 5 mg of amlodipine per day for 4 weeks. Up-titration to eplerenone 50 mg and amlodipine 10 mg for an additional 4 weeks.
3. Obtain basal metabolic rate, cardiac output and other indices of cardiac performance, cognitive abilities, and rating of depression and anxiety symptoms at baseline and after 8 weeks of treatment.
4. Obtain blood pressure measures at all visits.
5. Obtain mood ratings at all visits.
6. Compare basal metabolic rate, cardiac output and other indices of cardiac performance between treatment groups.
7. Compare difference in SBP and DBP between treatment groups.
8. Compare differences in plasma insulin, serum electrolytes, plasma renin activity, cortisol and aldosterone concentrations, urinary albumin excretion, and glomerular filtration rate between treatment groups.
9. Compare mood rating as well as symptoms of depression and anxiety between treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure (SBP) between 140 and 160 mmHg and/or a diastolic blood pressure between 90 and 100 mmHg who also have a body mass index > 30-45.
* Women must be post menopausal

Exclusion Criteria:

* Women of child bearing potential
* BMI less than 30 or greater than 45
* A creatinine > 1.8 for females and > 2.0 for males
* Type 1 or type 2 diabetes
* Current evidence of alcohol or drug abuse problems

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Basal metabolic rate | Pre and post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marion Wofford, MD, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- The University of Mississippi Clinical Research Program, Jackson, Mississippi, United States